CLINICAL TRIAL: NCT07372482
Title: Evaluating the Impact of Fat and Sugar Replacer Blends on Gastrointestinal Tolerance in Biscuits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: KBE073 / INQ-2405
Record Dates: First submitted 2025-07-23; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Tolerance; Healthy Population
Keywords: sugar replacers; fat replacer; gastrointestinal symptoms; Bowel Habits - Bristol Stool Scale (BHD-BSS); Gastrointestinal Tolerance Questionnaire (GITQ); Acute; Biscuits
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Intervention Model Description: In a 7-way cross-over, 14 sequences are required to obtain a balanced design. Orders will be assigned to participants in the order they attended for the first visit after being recruited. Four of these sequences will be separately randomized to create n=56 random sequences. If more subjects are recruited to replace drop-outs then the first new recruit will be assigned the sequence assigned the first drop-out, the second new recruit to sequence assigned to the second drop-out, etc.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The products will be labelled with a code, and participants will not be informed which test meal is which. Double blinding will be achieved by identifying the treatments by code on the case report forms and, in the database, so that those doing the statistical analysis and the study sponsor will be unaware of the treatment assignments. After the database has been created, cleaned, and locked a copy will be sent to the sponsor and then the codes will be broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control biscuit (Placebo Comparator): Sandwiched biscuit with usual sugar and fat content (2 servings = 60g)
  Interventions: Other: Control sandwiched biscuit with sugar
- Control biscuit reduced in fat with EPG (Active Comparator): Sandwiched biscuit with usual sugar content and fat partly replaced by EPG in basecake (2 servings = 60g)
  Interventions: Other: Test sandwiched biscuits with creme
- Sugar reduced biscuit with blend 1 (Active Comparator): Sandwiched biscuit reduced in sugar and containing sugar-replacer blend 1 (2 servings = 60g)
  Interventions: Other: Test sandwiched biscuits with creme
- Sugar reduced biscuit with blend 1 + EPG in basecake (Active Comparator): Sandwiched biscuit reduced in sugar and containing sugar-replacer blend 1 and EPG replacing fat in basecake (2 servings = 60g)
  Interventions: Other: Test sandwiched biscuits with creme
- Sugar reduced biscuit with blend 1 + EPG in basecake & creme (Active Comparator): Sandwiched biscuit reduced in sugar and containing sugar-replacer blend 1 and EPG replacing fat in basecake & creme (2 servings = 60g)
  Interventions: Other: Test sandwiched biscuits with creme
- Sugar reduced biscuit with blend 2 (Active Comparator): Sandwiched biscuit reduced in sugar and containing sugar-replacer blend 2 (2 servings = 60g)
  Interventions: Other: Test sandwiched biscuits with creme
- Sugar reduced biscuit with blend 2 + EPG in basecake (Active Comparator): Sandwiched biscuit reduced in sugar and containing sugar-replacer blend 2 and EPG replacing fat in basecake (2 servings = 60g)
  Interventions: Other: Test sandwiched biscuits with creme

INTERVENTIONS:
Other: Test sandwiched biscuits with creme — Acute intake
  Arms: Control biscuit reduced in fat with EPG; Sugar reduced biscuit with blend 1; Sugar reduced biscuit with blend 1 + EPG in basecake; Sugar reduced biscuit with blend 1 + EPG in basecake & creme; Sugar reduced biscuit with blend 2; Sugar reduced biscuit with blend 2 + EPG in basecake
Other: Control sandwiched biscuit with sugar — Acute intake
  Arms: Control biscuit

SUMMARY:
This study is a randomized, double-blind, crossover trial aiming at evaluating the gastrointestinal tolerance and bowel habits of sugar- and fat- replacer ingredients and blends (maltitol, polydextrose, allulose and EPG)

DETAILED DESCRIPTION:
The study will have a randomized, double-blind, crossover design with 8 visits consisting of one screening visit and 7 study visits (3 to 14-day interval between the start of each visit) across 4-12 weeks. Participants will be randomized to a test sequence and, during the course of the study, will complete 7 trial arms. At each visit eligible participants will come to INQUIS between 8-11am, and ~1-2h after consuming their usual breakfast at home. After rating the severity of GI symptoms, participants will consume one of the investigational products with a drink of water (250ml) and then be free to leave. The severity of 11 symptoms will be rated at 0, 2, 4, 6, 10 and 24h: Abdominal bloating, Abdominal pain, Gas/flatulence, Gas with discharge, Burping, Reflux (heartburn), Stomach rumbling (borborygmus), Urgency of bowel movement, Oily spotting (leakage), Nausea and Vomiting. The severity of each symptom will be rated by the subject as None, Mild, Moderate or Severe (these ratings will be assigned scores of 0, 1, 2 or 3, respectively). For each bowel movement (BM) passed during the 24h period, participants will be asked to record: the time, if they had to strain (yes or no), if they experienced discomfort (yes or no), if they felt there was incomplete evacuation (yes or no), if they had oily evacuation (oil separated from the stools) (yes or no), if they had oily stool (oily lumps in the stool) (yes or no) and the consistency of the stool rated using the using the Bristol Stool Scale (BSS).

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating, healthy individuals aged 18-55 years, inclusive
* Body Mass Index (BMI) 18.5-32.0kg/m², inclusive
* No major illness, trauma or surgery requiring hospitalization within 3 months of the screening visit
* Ability to understand the study procedures and willing to provide informed consent to participate in the study
* Non-smokers or smokers who smoke <10 cigarettes/day and are willing not to change nicotine habits during the study period
* Willing to limit alcohol consumption to ≤3 standard drinks/day and ≤7 standard drinks/week during the study period
* Willing to refrain from any marijuana or hemp products during the study period
* Normal bowel habits (>2 bowel movements/week and <3 bowel movements per day)
* Consumes ≤4 servings/day of fruits and vegetables combined and ≤3 (women) or ≤4 (men) servings/day of whole grains using the definitions of "serving" .
* Participants must have a cell phone/tablet/computer and be willing and able to use it to collect study data
* Participants must be eligible to receive income in Canada and be covered by a health insurance plan such as OHIP (Ontario Health Insurance Plan)
* Participants are willing to follow current COVID guidelines with respect to attending study visits

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Chronic moderate to severe gastrointestinal symptoms
* Use of systemic antibiotics, antifungals or antiparasitics in the past 3 months and during the experimental period
* Use of medications, supplements, and products which may affect the results (laxative, anti-diarrhea, anti-constipation drugs, high fiber supplements)
* Individuals with any medical conditions or use of supplements or medications that increase risk to the subject or others or may affect the results, as judged by the Principal - Investigator
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS safety guidelines
* Known intolerance, sensitivity, or allergy to any ingredients in the study test products
* Subject is currently participating or recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement, or lifestyle modification

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Total Area Under the Curve (tAUC) of composite gastrointestinal Symptom score | tAUC between 0 and 24 hours
  total area under the curve (tAUC) of the composite GastroIntestinal symptom score (sum of the scores for the 11 GI symptoms). The score values can range from 0 up to 24 with the higher values showing the higher levels of symptoms (worse conditions).

SECONDARY OUTCOMES:
Total Area Under the Curve of each individual gastrointestinal symptom | tAUC between 0 and 24 hours
  Total Area Under the Curve of each of the individual 11 gastrointestinal symptoms (Abdominal bloating, Abdominal pain, Gas/flatulence, Gas with discharge, Burping, Reflux (heartburn), Stomach rumbling (borborygmus), Urgency of bowel movement, Oily spotting (leakage), Nausea and Vomiting). Each symptom range from 0 up to 3 with 3 showing the highest / worse condiiton of symptoms
Frequency of composite score > 1 at each time point | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants who have a composite GastoInestinal symptom score >1 (moderate-to-severe) at each time point. The composite score can range from 0 up to 24 with the higher values showing the higher levels of symptoms (worse conditions)
Frequency of Diarrhea within 24 hours | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants with diarrhea, defined as 3 or more type 6 or 7 stools (based on the BSS) within the 24 hour period after consumption of the study products
Time for maximum score for abdominal bloating | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score for bloating
Maximum score for abdominal bloating | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for abdominal bloating | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time of maximum score for abdominal pain | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for abdominal pain | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for abdominal pain | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for flatulence | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for flatulence | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for flatulence | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for gas with discharge | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for gas with discharge | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for gas with discharge | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for burping | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for burping | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for burping | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for reflux | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for reflux | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for reflux | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for stomach rumbling | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for stomach rumbling | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for stomach rumbling | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for Oily spotting (leakage) | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for Evaluation oily spotting (leakage) | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for oily spotting (leakage) | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for nausea | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for nausea | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for nausea | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Time for maximum score for vomiting | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Time of the maximum score
Maximum score for vomiting | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Proportion of participants reporting any (score>0) or moderate/severe (score >1) at each time point
Maximum score for vomiting | Evaluation performed at time 0, 2, 4, 6, 10 and 24 hours
  Maximum detected score (which can range from 0 up to 3)
Number of bowel movements | Evaluation performed over 24 hour after consumption of study products
  Number of bowel movements over the 24 hours
straining during bowel movement | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants having to strain or not
discomfort during bowel movement | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants having discomfort or not
incomplete evacuation | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants declaring incomplete evacuation or not
oily evacuation (oil separated from the stools) | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants declaring having oily evacuation (oil separated from the stools)
oily stool (oily lumps in the stool) | Evaluation performed over 24 hour after consumption of study products
  Proportion of participants declaring having oily stool (oily lumps in the stool)
Stool consistency based on bristol stool scale | Evaluation performed over 24 hour after consumption of study products
  mean stool consistency on Bristol Stool Scale (BSS). The scale provide values from 1 to 7 depending on the type of stool with 1 being the driest stools and 7 the most liquid one.

CONTACTS AND LOCATIONS:
Locations (1):
- Inquis Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No